CLINICAL TRIAL: NCT07315243
Title: Modified Amniotic Fluid Scoring Model Incorporating Fetal Bladder Assessment
Brief Title: Modified Amniotic Fluid Score With Fetal Bladder Assessment
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Salah Eldin Ali Hassan, Resident at Obstetrics and Gynecology Department, Assiut University, Assiut University
Other Study IDs: Modified Amniotic Fluid Score
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Amniotic Fluid Scoring Model; Fetal Bladder Assessment
Keywords: Modified Amniotic Fluid Scoring Model; Fetal Bladder Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study will prospectively enroll pregnant women with singleton pregnancies between 20 and 38 weeks of gestation who attend Assiut University Hospital for routine or indicated ultrasound assessment of amniotic fluid. The aim is to develop and validate a modified amniotic fluid scoring model that combines standard ultrasound measures of amniotic fluid volume with fetal bladder size and appearance. The study will compare the ability of this new scoring model to detect abnormal amniotic fluid volume against conventional ultrasound methods and will explore how fetal bladder measurements relate to amniotic fluid indices.

DETAILED DESCRIPTION:
This prospective observational cohort study will be conducted in the Obstetrics and Gynecology Department at Assiut University Hospital and will enroll 70 pregnant women aged 18-45 years with singleton pregnancies between 20 and 38 weeks of gestation who are referred for routine or clinically indicated ultrasound assessment of amniotic fluid volume. The study aims to develop and validate a modified amniotic fluid scoring model that integrates standard sonographic measures of amniotic fluid volume, including the amniotic fluid index and single deepest pocket, with predefined fetal bladder parameters such as bladder presence, morphology, and longitudinal and transverse diameters measured at maximal filling.

Eligible participants will undergo a standardized ultrasound examination using a high-resolution machine with a curvilinear transducer; the uterus will be systematically scanned to obtain AFI and single deepest pocket measurements, followed by a dedicated five-minute assessment of the fetal bladder to document its size, appearance, and any observed micturition events. All sonographic assessments will be performed by experienced sonographers following uniform protocols, and approximately 10 percent of examinations will be re-scanned by a second sonographer to assess interobserver reliability, with images and measurements digitally archived for blinded review.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 18-45 years.
* Singleton pregnancy between 20 and 38 weeks of gestation.
* Women attending Assiut University Hospital for routine or indicated ultrasound assessment of amniotic fluid volume.
* No known major fetal anomalies at the time of inclusion.
* Able and willing to provide written informed consent.

Exclusion Criteria:

* Multiple pregnancy (e.g., twins, triplets).
* Pregnancies with known chromosomal or major structural fetal anomalies diagnosed prior to enrollment.
* Maternal systemic diseases known to affect amniotic fluid volume (e.g., pregestational or gestational diabetes, chronic hypertension, renal disease).
* Contraindications to ultrasound examination.
* Inability to provide informed consent or anticipated poor compliance with study procedures.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: Pregnant women aged 18-45 years with singleton pregnancies between 20 and 38 weeks of gestation attending the Obstetrics and Gynecology Department at Assiut University Hospital for routine or indicated ultrasound assessment of amniotic fluid volume.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Sensitivity Of The Modified Amniotic Fluid Scoring Model | At the index obstetric ultrasound examination during pregnancy (single visit per participant).
  Proportion of pregnancies with abnormal amniotic fluid volume (oligohydramnios or polyhydramnios) correctly identified as abnormal by the modified amniotic fluid scoring model incorporating fetal bladder assessment, using conventional ultrasound assessment (AFI/SDP) as the reference standard.

SECONDARY OUTCOMES:
Correlation Between Fetal Bladder Size And Amniotic Fluid Volume | At the same index obstetric ultrasound examination during pregnancy (single visit per participant).
  Correlation coefficient between fetal bladder dimensions (longitudinal and transverse diameters measured at maximal filling) and amniotic fluid volume indices (AFI and single deepest pocket) to assess the relationship between bladder size and amniotic fluid volume.